CLINICAL TRIAL: NCT06933173
Title: Mind-Body in Long COVID and Myalgic Encephalomyelitis Study (MILES): A Patient-Centred RCT
Brief Title: RCT of Mind-body in Long COVID and Myalgic Encephalomyelitis
Acronym: MILES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: College of Physicians and Surgeons of Alberta (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00138185
Record Dates: First submitted 2025-04-15; First posted 2025-04-18 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Myalgic Encephalomyelitis/Chronic Fatigue Syndrome
Keywords: Myalgic encephalomyelitis/Chronic fatigue syndrome; Mind-body intervention; Long COVID; RCT; Patient engagement
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Post-Acute COVID-19 Syndrome; Patient Participation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DNRS intervention group (Experimental)
  Interventions: Other: Dynamic neural retraining system
- Wait-list control group (No Intervention): The waitlist control group will complete the experimental intervention after 4 months. During the waiting period, they will continue to receive usual care and will be asked to not participate in any other new treatments.

INTERVENTIONS:
Other: Dynamic neural retraining system — Description: The DNRS program includes the following components: 1) cognitive-behavioural therapy; 2) mindfulness-based cognitive restructuring; 3) emotional restructuring therapy; 4) neural linguistic programming; 5) incremental training; and 6) behaviour modification therapy. DNRS offered in this study includes a 14-hour online course followed by a 12-week online "LIVING DNRS" group support program. The 14-hour online course includes a variety of exercises, instructional videos, and a workbook. Upon completion, participants are offered a 12-week LIVING DNRS Group Support program which provides individuals with support in how to best implement DNRS into their daily lives with the help of a trained facilitator as well as peer support.
  Arms: DNRS intervention group

SUMMARY:
We are studying the effect of a mind-body treatment for people with Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) with or without Long COVID (LC). Our team recognizes that ME/CFS and Long COVID are serious, debilitating, biomedical conditions.

ME/CFS can affect many different parts of the body, such as the nervous system, immune system, and metabolism. It is hypothesized that central sensitization (i.e., when nerves get too excited) may influence these complex conditions and may make symptoms worse.

This study explores a mind-body program called the Dynamic Neural Retraining System™, or DNRS™.

Mind-body interventions (MBIs) focus on how the brain, mind, body, and behaviour interact to improve health and well-being. These techniques help people become more aware of themselves, take better care of their health, and boost mood, quality of life, and coping skills. MBIs use the brain's ability to change (neuroplasticity) by reinforcing certain thoughts, feelings, or behaviours that support changes in biology and function. MBIs may influence physical health by affecting how the brain and body communicate through chemicals such as hormones and neurotransmitters. Objective fMRI evidence shows that practising MBIs can change brain structure and function. This makes MBIs a potential good fit for people with chronic illnesses like ME/CFS and LC, which involve complex interactions between the brain, immune system, and hormones.

There is no rigorous peer-reviewed evidence that DNRS is effective. Our study will address this question using subjective and objective measurements in a multiple-methods wait-list randomized controlled trial.

The objectives of this study are to: 1) examine the effectiveness of the DNRS program for individuals diagnosed with ME/CFS with and without Long COVID, compared to a treatment-as-usual wait-list control group on a range of patient-reported outcomes including health-related quality of life, fatigue, pain, anxiety and depression and objective measures including daily steps, heart rate variability, and sleep; 2) quantify metabolic changes through untargeted serum metabolomics profiling, 3) determine if metabolomics screening can predict treatment responsiveness to DNRS; and 4) identify the microbial signatures of large bowel microbiota in Long COVID patients pre and post MBI.

A descriptive qualitative study will also be conducted in a sample of participants to learn more about their experiences during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older;
* Individuals diagnosed with ME/CFS, according to the Institute of Medicine (2015) criteria, for more than six months.

Exclusion Criteria:

Individuals who: 1) are too ill to participate; 2) lack reliable internet; 3) cannot communicate in English; 4) Presently have or ever had inflammatory bowel disease; and/or 5) Have been prescribed or used an oral or systemic (infusion) antibiotic in the past one month-;; 6) are participating in a concurrent study; 7) are participating in a concurrent mind-body intervention during the study period including

* Art Therapy
* Autogenic training
* Biofeedback/neurofeedback
* Breathing exercise
* Cognitive restructuring
* Dynamic Neural Retraining System
* Emotional Freedom Techniques (EFT)
* Eye movement desensitization and reprocessing (EMDR)
* Guided imagery
* Hypnotherapy/self-hypnosis
* Meditation (mindfulness, mantra, guided, transcendental)
* Mindfulness-based cognitive therapy (MBCT)
* Mindfulness-based Stress Reduction (MBSR)
* Music therapy
* Neurolinguistic programming
* Psychological flexibility
* Qigong
* Relaxation therapy (relaxation response, progressive muscle relaxation)
* Tai Chi
* Visualization
* Yoga and/or starting any other new treatment during the study period, including any mind-body therapy, psychotherapy, prescription medication, over-the-counter medication, etc; 8) have any active medical condition (untreated/uncontrolled) that may explain the presence of fatigue including:
* untreated hypothyroidism (including Hashimoto's disease)
* hyperthyroidism
* diabetes mellitus
* iron deficiency anemia
* other treatable anemia
* iron overload syndrome
* adrenal insufficiency
* Cushing's syndrome
* anorexia nervosa
* iatrogenic conditions such as side effects or interactions of medication(s) or supplements

  • Rheumatological disorders:
* rheumatoid arthritis
* lupus
* polymyositis
* polymyalgia rheumatica
* Sjogren's Syndrome
* Ehlers Danlos Syndromes [Hypermobility type]

  • Other heritable disorders of connective tissue:
* Marfan syndrome
* Stickler syndrome etc.

  * Multiple sclerosis
  * Celiac disease
* Note: Patients with celiac disease can present without gastrointestinal symptoms

  • Immune disorders
* such as HIV/AIDS

  • Sleep disorders
* including obstructive sleep apnea

  • Prior illnesses may relapse or may not have completely resolved during treatment.
* Examples are certain malignancies
* leukemia
* infectious diseases such as tuberculosis and chronic hepatitis

  • Active primary psychiatric disorders
* eating disorders
* alcohol
* substance use disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Physical functioning | Difference in changes from baseline to post intervention/post waiting (within 4 weeks of completing the DNRS program or waiting period)
  Physical functioning of health-related quality of life (HRQL) as measured by the Short Form 36-item Health Survey (SF-36) (V1)

CONTACTS AND LOCATIONS:
Overall Officials: Sunita Vohra, MD MSc FRCPC FCAHS, Principal Investigator — University of Alberta; Eleanor Stein, MD FRCPC, Principal Investigator — University of Calgary
Locations (3):
- Canada (3):
  - Peter Lougheed Hospital, Calgary, Alberta
  - University of Alberta Hospital/Kaye Edmonton Clinic, Edmonton, Alberta
  - Women's College Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided